CLINICAL TRIAL: NCT02977728
Title: Olfactory Function in Patients With Acute Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Hôpital de Viege (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01442
Record Dates: First submitted 2016-11-17; First posted 2016-11-30 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Mild Traumatic Brain Injury
Keywords: MTBI; olfaction; acute
MeSH Terms: conditions — Brain Concussion; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mild Traumatic Brain Injury: The investigators will include patients who have been diagnosed with a mild traumatic brain injury (Glasgow Coma Scale 13 and above). The patients will be aged between 18 and 55 years old and admitted to the Hospital Visp in the 24 hours preceding the testing.
  Interventions: Other: Olfactory Evaluation
- Orthopaedic Injury: The investigators will include patients who have been diagnosed with a traumatic orthopedic injury to one of their limbs. The patients will be aged between 18 and 55 years old and admitted to the Hospital Visp in the 24 hours preceding the testing.
  Interventions: Other: Olfactory Evaluation

INTERVENTIONS:
Other: Olfactory Evaluation — The investigators will evaluate the olfactory system of all participants by the use of the Sniffin'Sticks batterie

SUMMARY:
In this project the investigators aim to evaluate olfactory and non-olfactory function in patients within the first 24h following a mild traumatic brain injury (acute mTBI) and compare their results to a group of age and sex matched control patients suffering from an orthopedic injury 24h prior to testing. The investigators then aim to follow them up 1 year after the trauma

DETAILED DESCRIPTION:
This is a research project in which health-related personal data is collected; the investigators will use coded data. Further this project is a cross-sectional study.

Procedure Potential participants will be identified via the collaborating physicians who will inquire about the interest of the patient to participate. The investigators will then approach patients in their room and inform them about the study. If the patient is interested they will sign the consent form and be included in the study.

Session 1: Session 1 will be carried out directly after inclusion into the study. First the investigators will execute olfactory tests subjective olfactory impairment, Sniffin' Sticks test (threshold, discrimination, identification) and subjective odor evaluation. This will approximately last one hour (with breaks). Participants will then have a break of 15-60 minutes. In the following the investigators will carry out the non-olfactory tests; this will last another 45 minutes.

Session 2: During inclusion, participants will be asked to give their contact details (email and postal address). 10 months after the first session, the investigators will contact them by email. The investigators will then send them a booklet of the UPSIT by mail. Participants will be asked to fill out the test and send it back with a prepaid envelope.

Recruitment Potential participants will be identified via the collaborating physicians who will inquire about the interest of the patient to participate. The investigators will then approach patients in their room and inform them about the study. If the patient is interested they will sign the consent form and be included in the study. Specifically, the responsible researcher will perform consecutive ongoing recruitment through daily clinical practice. The investigators will also carry out the screening.

Criteria for withdrawal / discontinuation of participants:

The participant participation in this study is strictly voluntary. They may refuse to participate or may discontinue their participation at any time without explanation, and without penalty or loss of benefits to which they are otherwise entitled. If they decide not to participate, or if they discontinue their participation, they will suffer no prejudice regarding medical care or their participation in any other research studies. They will be informed of any new findings that may affect their willingness to continue their participation.

The study doctor may end the participant participation for administrative reasons unrelated to the purpose of the study. In addition, the Swiss Ethics Committees on research involving humans may terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will include patients aged between 18 and 55 years old
* admitted to the Hospital Visp in the 24 hours preceding the testing
* MTBI group: The investigators will include patients who have been diagnosed with a mild traumatic brain injury (Glasgow Coma Scale 13 and above) within 24h before inclusion.
* Orthopaedic Group: The investigators will include patients who have been diagnosed with a traumatic orthopaedic injury to one of their limbs within 24 hours before inclusion.

Exclusion Criteria:

* are under the influence of alcohol or drugs during the time of testing
* patients with a known history of traumatic brain injury (e.g., a prior concussion)
* patients with a known and pharmacologically treated neurological or psychiatric diseases
* patients who have suffered from an injury to the face (such as a broken nose)
* patients who do not have German, French or English as their first language
* For the orthopaedic group : The investigators will exclude patients who, in addition to their orthopaedic trauma, have suffered from a brain injury due to their trauma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The investigators will include a total of 30 patients with acute (into the first 24 hours) mild TBI and the same number of patients with an orthopaedic injury not involving the head.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the objective and subjective olfactory function in patients following an acute mild traumatic brain injury | The investigators will evaluate the olfactory system within 24h following the trauma
  The investigatos will assess several different aspects of olfactory function with the Sniffin' Sticks test.Threshold: At each trial 3 pens are presented in a randomized order, two of which contain the solvent and one the odorant at a certain dilution. The subjects' task is to detect the odour-containing pen.Discrimination: Odour discrimination will be assessed by presenting triplets of pens in a randomized order. Two of them contain the same odorant, while the third contains a different odorant. Subjects have to determine which of the three odour- containing pens smells different. Identification: Odour identification will be assessed by means of common odours, presented in 16 different sticks. Using a forced choice approach, participants will select the best descriptor from a list of four for each odorant.Subjective olfactory impairment:The investigators will use an adapted version of the Questionnaire of Olfactory Disorders to determine the changes in olfactory function.

SECONDARY OUTCOMES:
Evaluate the anxiety levels in patients following an acute mild traumatic brain injury | The investigators will evaluate the anxiety levels within 24h following the trauma
  The investigators will assess anxiety levels by using the Hospital Anxiety and Depression Scale (HADS). The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depressionAlso, the Hamilton Anxiety Rating Scale, a 14-item scale designed to assess anxiety severity, will be administered by the examiner. It has been suggested to reflect subclinical expression of anxiety disorders.
Evaluate the cognitive profil of the patients following an acute mild traumatic brain injury | The investigators will evaluate the cognitive profils within 24h following the trauma
  The Trail Making Test version A and B will be use in order to evaluate visual attention and task switching. This test consists of connecting dots carrying numbers and letters. We will further use the Stroop test to evaluate inhibition and interference in our participants. In addition we will use the Digit symbol substitution test, which measures speed of information processing. Finally, we will assess working memory, attention and mental control by using the letter number sequencing portion of the WAIS. All these tests have been shown to be sensitive to TBI. We will further evaluate cognitive impairment by means of the RBANS (Repeatable Battery for the Assessment of Neuropsychological Status). Offering valuable enhancements, the RBANS Update provides a brief, individually administered battery to measure the general cognitive profil.
Evaluate the post-concussion symptoms in patients following an acute mild traumatic brain injury | The investigators will evaluate the post-concussion symptoms within 24h following the trauma
  The investigators will use the Rivermead post-concussion symptoms questionnaire. It allows for determining the presence and severity of 16 post-concussion symptoms including somatic, cognitive and emotional symptoms
Evaluate the olfactory system one year post-tbi by the use of the UPSIT | One year after the mild traumatic brain Injury
  The investigators will send by mail the UPSIT: The University of Pennsylvania Smell Identification Test (UPSIT) one year post-injury. The UPSIT is a "scratch and sniff" test based on microencapsulated odorants which are released from the surface of strips by means of a pencil. The patient is asked to choose 40 odorants on a multiple-choice list comprising four items each.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Frasnelli, Ph.D., Study Director — Sacre-Coeur Hospital

IPD SHARING:
Plan to Share IPD: No